CLINICAL TRIAL: NCT05827211
Title: Asepsis During Periodontal Surgery Involving Oral Implants and the Usefulness of Antibiotics: a Prospective, Randomized, Controlled Clinical Trial
Brief Title: The Usefulness of Antibiotics in Smokers Receiving Dental Implants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Arab American University (Palestine) (Other)
Responsible Party: Principal Investigator, Mahmoud Abu-Ta'a, Associate Professor, Arab American University (Palestine)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: Antibiotics
Record Dates: First submitted 2023-03-31; First posted 2023-04-24 (Actual); Last update posted 2023-07-20 (Actual); Status verified 2023-07

CONDITIONS: Dental Implant Therapy
MeSH Terms: interventions — Anti-Bacterial Agents

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test group (Experimental): Participants in this group will receive Doxycycline 200 mg 1 h pre-op and 100 mg for 9 days post-op in combination with dental implant therapy.
  Interventions: Procedure: Antibiotic group
- Control group (Placebo Comparator): Participants in this group will receive a placebo 200 mg 1 h pre-op and 100 mg for 9 days post-op in combination with dental implant therapy.
  Interventions: Procedure: Non-Antibiotic group

INTERVENTIONS:
Procedure: Antibiotic group — Partially or fully edentulous smoker patients will be treated by dental implants and will receive systemic antibiotics
  Other Names: Dental implant insertion + Antibiotics
  Arms: Test group
Procedure: Non-Antibiotic group — Partially or fully edentulous smoker patients will be treated by dental implants and will receive placebo
  Other Names: Dental implant insertion + Placebo
  Arms: Control group

SUMMARY:
Objectives: This randomized clinical trial will compare the usefulness of pre- and postoperative antibiotics while strict asepsis will be followed during periodontal surgery in smokers diagnosed with Stage III Grade C Generalized Periodontitis.

Material and Methods: Two groups of 40 consecutive patients each with fully or partially edentulous jaws will be enrolled. Antibiotics group (GrAB+): will receive oral doxycycline 200 mg, 1 h pre-operatively and 100 mg g for 9 days post-operatively. Non-antibiotics group (GrAB- ): will receive a placebo (no antibiotics). Bacterial samples will be taken from the peri-oral skin before and at the end of the surgery. In 12 patients in each group, samples will also be taken from the nares. A visual analogue scale will evaluate symptoms of infection/ inflammation by both the patient and the periodontist at suture removal.

ELIGIBILITY:
Inclusion Criteria:

* smoker
* in need of dental implant therapy
* above 18 years of age

Exclusion Criteria:

* allergy to doxycycline,
* need for endocarditis prophylaxis,
* any systemic or local immunodeficiency,
* uncontrolled diabetes mellitus,
* previous radiation therapy in the head and neck area

Ages: 19 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2023-04-02 (Actual); Primary Completion 2023-04-30 (Actual); Study Completion 2023-06-10 (Actual)

PRIMARY OUTCOMES:
Rate of post-operative infection | 7 days
  signs of infection (fever > 38 degrees celsius, spontaneous bleeding, pus, swelling, etc.) post-operatively will be checked at suture removal

CONTACTS AND LOCATIONS:
Overall Officials: Mahmoud Abu-Ta'a, Principal Investigator — Department of Dental sciences, Faculty of Graduate Studies, Arab American University (AAUP)
Locations (1):
- Mahmoud Abu-Ta'a, Ramallah, Palestinian Territories

IPD SHARING:
Plan to Share IPD: Undecided